CLINICAL TRIAL: NCT02203383
Title: Sleep Disordered Breathing in Patients With Implanted Cardiac Devices: Assessment of the Change in Sensitivity to Carbon Dioxide With Cardiac Resynchronization Therapy.
Brief Title: The Effect of CRT on the Hypercapnic Ventilatory Response
Status: Suspended | Type: Observational
Why Stopped: Pending further equipment and staff
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 14/LO/0078
Record Dates: First submitted 2014-07-28; First posted 2014-07-29 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-11

CONDITIONS: Sleep Disordered Breathing; Heart Failure
Keywords: Cardiac Resynchronization Therapy; Central Sleep Apnoea; Sleep Disordered Breathing; Heart Failure; Hypercapnic Ventilatory Response
MeSH Terms: conditions — Sleep Apnea Syndromes; Heart Failure; Sleep Apnea, Central

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Pts with CSA for CRT implantation: Patients with heart failure (EF<40%) and moderate to severe CSA (>15 events per hour, >50% Central)
  Interventions: Device: CRT Implantation
- No Sleep Apnoea for CRT implantation: Heart failure (EF < 40%) but no significant sleep apnoea (<5 events per hour).
  Interventions: Device: CRT Implantation

INTERVENTIONS:
Device: CRT Implantation — Implantation of a biventricular pacemaker or defibrillator.
  Other Names: INVIVE; INCEPTA; AUTOGEN

SUMMARY:
Central Sleep Apnoea (CSA) affects up to half of patients with severe heart failure and is associated with a poor prognosis. CSA is manifest as episodes of deep breathing interspersed with very shallow or absent breathing and is largely due to an exaggerated response to rising carbon dioxide in the blood, which normally drives how hard we breathe. Cardiac Resynchronization therapy (CRT), in which a pacemaker is implanted to improve co-ordinated contraction of the heart, has been shown to reduce the severity of CSA in some patient groups. We aim to determine whether this improvement is due to normalization of the body's response to carbon dioxide in the blood. Our hypothesis is that CRT improves CSA by normalizing the brain's response to carbon dioxide.

DETAILED DESCRIPTION:
Sleep disordered Breathing is common in heart failure, affecting around half of patients. This may be Obstructive Sleep Apnoea due to loss of pharyngeal muscle tone (OSA, associated with obesity and snoring and predisposing to hypertension, heart attack and stroke) or Central Sleep Apnoea (CSA). CSA is particularly prevalent in severe heart failure and associated with an adverse prognosis. The mechanism involves reflex hyperventilation due to pulmonary oedema, exaggerated chemosensor response to hypercapnoea associated with increased sympathetic nervous system activation and a prolonged circulation time.

It is known that CRT improved CSA in 'responders' but the mechanism is unknown. We hypothesis that CRT normalizes the respiratory response to carbon dioxide (the hypercapnic ventilatory response - HCVR).

We will screen patients undergoing CRT with an Embletta sleep study to identify a group with moderate to severe CSA and a group with no sleep apnoea (controls). Patients will undergo assessment of the hypercapnic ventilatory response with a Read Re-Breathe test prior to device implantation and 6 weeks and 6 months afterwards. The gradient of minute ventilation vs PaCO2 will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure with reduced ejection fraction (<40%)
* Either no significant sleep disordered breathing or moderate to severe CSA
* Able to consent to the study
* Ambulatory
* Aged 18-100 years

Exclusion Criteria:

* Patients on Non-Invasive Ventilation
* Predominant OSA
* Unable to consent or attend for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with heart failure with reduced ejection fraction (<40% on echocardiography) due to undergo implantation of a biventricular pacemaker, with either no significant sleep disordered breathing or moderate to severe CSA.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2014-06; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
The change in gradient of minute ventilation vs end tidal CO2 before and after CRT (the hypercapnic ventilatory response). | 6 weeks and 6 months

SECONDARY OUTCOMES:
6 minute walk distance | 6 weeks and 6 months
Change in resting PaCO2 | 6 weeks and 6 months
Change in left ventricular ejection fraction | 6 weeks and 6 months
Change in plasma B-Type Natriuretic Peptide level | 6 weeks and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ali Vazir, PhD, Principal Investigator — Imperial College. Royal Brompton Hospital; Martin Cowie, MD, Study Chair — Imperial College London
Locations (1):
- Royal Brompton and Harefield NHS Foundation Trust, London, United Kingdom